CLINICAL TRIAL: NCT05765409
Title: Assessment of the Effectiveness of an Integrative Therapy for Cannabis Misuse in Adolescents (Randomized Controlled Trial of Non-inferiority)
Brief Title: Assessment of the Effectiveness of an Integrative Therapy for Cannabis Misuse in Adolescents
Acronym: TIMCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D22-P019
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Cannabis Use Disorder
Keywords: Randomized Controlled Trial; Cannabis Use Disorder; Adolescents; Young adults; Motivational Interviewing; Cognitive and Behavioral Therapy; Attachment-based Intervention
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This will be a single-blinded, randomised, comparative therapeutic interventions, controlled trial.
  This is a prospective, randomized, single-blind, two-arm, parallel, multicenter study to evaluate the non-inferiority of an Integrative Therapy for Adolescent Cannabis Misuse (TIMCA) compared to the Treatment As Usual (TAU) control group using an Adaptive Group-Sequential non Inferiority Study Design. Two interim analyses are planned (when 30 and 60 subjects have completed the study).
  Both interventions will take place under similar conditions: 10 sessions, once a week, delivered by clinical psychologists who will be supervised.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIMCA (Experimental): The intervention will combine elements of motivational interviewing, cognitive and behavioral therapy and an attachment-based intervention. Sessions with both the adolescent and his parents are planned.
  Interventions: Other: TIMCA
- Treatment as Usual (Active Comparator): The comparator, an active control, will be Treatment As Usual" (TAU) group, i.e., the therapy usually practiced in the services. Given the multiplicity of investigating centers and the different treatments offered according to the patient's problems, it seems difficult to choose a single reference treatment for the control arm. Each investigating center undertakes to adopt the treatment that seems most effective and appropriate for each patient
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: TIMCA — TIMCA is an individual therapy that will include the parents at certain points in the therapy .
  It will consist of two sessions of MI, two sessions of CBT, five sessions of ABI and one final session of summary to conclude the therapy.
  Out of 10 sessions, there will be three with the parents and the adolescent together.
  Arms: TIMCA
Other: Treatment as Usual — TAU will consist of several approaches including analytical, cognitive-behavioral , intepersonal psychotherapy.
  Each therapist will be asked to specify the approach used as well as the therapeutic axes.
  Arms: Treatment as Usual

SUMMARY:
The primary objective of this study is to evaluate an Integrative Therapy for Adolescent Cannabis Use (TIMCA), integrating elements of Motivational Interviewing (MI), Cognitive Behavioral Therapies (CBT) and an Attachment-Based Intervention (ABI), (IBA),compared to Treatment As Usual (TAU) on cannabis use.

The secondary objectives of the study are:

To assess the effectiveness of the TIMCA, in comparison to the TAU, on: (1) Relationship quality with parents, (2) Relationship quality with closest friend, (3) Emotional regulation strategies, (4) Depressive symptomatology, (5) Anxiety symptomatology, (6) Adherence to therapy

DETAILED DESCRIPTION:
Cannabis is the most used psychoactive substance in the world after tobacco and alcohol, particularly among adolescents and young adults. Cannabis use during adolescence can lead to cognitive, psychological, academic, and social consequences, causing significant distress. In 2019, French adolescents reported one of the highest levels of cannabis experimentation and use (past month) in Europe (5th and 2nd respectively) (Philippon & Spilka, 2020). Regular use of cannabis during adolescence can cause or reinforce psychological suffering in both the young person and those around him/her, and therefore constitutes a major public health issue. Although psychotherapeutic techniques form the basis of treatment for Cannabis Use Disorder (CUD), relapse is common at the follow-up assessment after therapy has ended (Gates et al., 2016; Walther et al., 2016). The literature shows the effectiveness of Motivational Interviewing (MI) on the one hand, and psychotherapies such as Cognitive Behavioral Therapies (CBT) and Multidimensional Family Therapy (MDFT) on the other. The most consistent and coherent evidence supports the combination of CBT and MI to decrease the frequency and severity of cannabis use. As the combination of MI and CBT has proven to be effective with young users, it seems important to add an Attachment-Based Intervention (ABI), as difficulties with interpersonal relationships and emotional regulation are risk factors for the development and maintenance of addiction in adolescents (Fairbairn et al., 2018; Rahioui, 2016).

This randomized, single-blind, two-arm, parallel, multicenter trial postulates that participants in the TIMCA group will have better outcomes than those in the Treatment As Usual (TAU) group in terms of cannabis use, quality of relationship with others, emotional regulation strategies, as well as anxiety-depressive symptomatology (during therapy, at the end of therapy, and at four weeks after the end of therapy).

ELIGIBILITY:
Inclusion Criteria:

* Aged 14 to 19 years 11 months 29 (or 30) days at the time of the inclusion visit
* Consulting as an outpatient center:
* Fulfilling the criteria for Cannabis Use Disorder (CUD) according to DSM 5 criteria (mild, moderate or severe)
* Fluent in oral and written French
* Benefiting from a social security plan
* Having signed their consent to participate (and their legal representative if applicable).

Exclusion Criteria:

* With an acute psychiatric disorder and/or a psychotropic treatment (a characterized depressive episode, a bipolar disorder, a psychotic disorder)
* With a substance use disorder other than cannabis and tobacco,
* Already engaged in another form of therapy
* Pregnant women at the time of inclusion
* Participants of age subject to a legal protection measure or unable to express their consent

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-06-09 (Estimated); Study Completion 2025-06-09 (Estimated)

PRIMARY OUTCOMES:
Cannabis use | 4 weeks after the end of treatment
  Cannabis use will be assessed via the TimeLine Follow Back (TLFB) (Robinson et al., 2014) and a urinanalysis (NarcoCheck)

SECONDARY OUTCOMES:
Parent and peer attachment | 4 weeks after the end of treatment
  Inventory of Parent and Peer attachment (IPPA) (Vignoli & Mallet, 2004)
Emotion regulation | 4 weeks after the end of treatment
  The Regulation of Emotions Questionnaire (REQ2) (Sequeira, 2013)
Anxiety symptomatology | 4 weeks after the end of treatment
  The Spielberger State-Trait Anxiety Inventory (STAI) (Spielberger et al., 1993)
Depressive symptomatology | 4 weeks after the end of treatment
  Beck Depression Inventory (BDI) (Byrne & Baron, 1994)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Rahioui, Doctor, Principal Investigator — GHU Paris Psychiatry & Neurosciences
Locations (1):
- GHU Paris Psychiatrie & Neurosciences, Paris, France